CLINICAL TRIAL: NCT03299452
Title: Clinical Studies by Using Alphacait to Screen Drug Combinations for Advanced Solid Tumor
Brief Title: Clinical Studies by Using Alphacait to Screen Drugs for Advanced Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haining Health-Coming Biotech Co., Ltd. (Other)
Collaborators: Alphacait, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alphacait 001
Record Dates: First submitted 2017-08-28; First posted 2017-10-03 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Cancer
Keywords: ex vivo high-throughput drug screening assay
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This single center, open-label, single arm, non-randomized study is designed to evaluate safety, progression-free survival(PFS),overall survival (OS), objective response rate (OPR), and disease control rate (DCR) of chemotherapy or target therapy or chinese medicine based on the Alphacait screening system in subjects with advanced malignant tumor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alphacait-guided therapy (Experimental): Drugs screened by the Alphacait screening system will be administered in accordance with the protocol of the drug specification or the CPSC guidelines until the patient progresses, intolerant, the patient withdrawn or the investigator determines that the medication must be discontinued.
  Interventions: Drug: Non Chemotherapy; Drug: Chemotherapy and target therapy; Drug: Chinese herb medicine

INTERVENTIONS:
Drug: Non Chemotherapy — Drugs screened by the Alphacait screening system will be administered in accordance with the protocol of the drug specification or the CPSC guidelines.
Drug: Chemotherapy and target therapy — Drugs screened by the Alphacait screening system will be administered in accordance with the protocol of the drug specification or the CPSC guidelines.
Drug: Chinese herb medicine — Drugs screened by the Alphacait screening system will be administered in accordance with the protocol of the drug specification or the CPSC guidelines.

SUMMARY:
This is a single-center, open-label, single-arm, non-randomized study designed to evaluate PFS, safety, overall survival (OS), objective response rate (OPR), disease control rate (DCR) and biomarkers of cancer therapy based on Alphacait screening system in subjects with advanced malignant tumor.

DETAILED DESCRIPTION:
Tumor heterogeneity leads to a significant difference in the rate of response to drugs in patients with the same pathological type. According to the information, the current initial effective rate of domestic and foreign chemotherapeutic single drug is no more than 30%, even if treated with repeated medication or replacement treatment program, the responsive rate is generally not more than 10%. This heterogeneity of tumor is the biological basis of precision medicine, and how to predict cancer drug sensitivity is a clinical need to solve the practical problems.

Traditional PDX (patient-derived engraft) technology utilizes patient's fresh tumor tissue (containing tumor cells, stromal cells and vascular components), and inoculates in immunodeficient mice to establish mouse tumor model. This method can better reflect the true biological characteristics of tumor, while the mouse tumor tissue can be continuously passed on, and greatly facilitate tumor biology research. According to the transplant site it can be divided into orthotopic transplantation and ectopic transplantation (mostly subcutaneous or renal transplantation). However, the traditional PDX model has its disadvantage of low success rate and time consuming. Most of the tumor matrix after transplantation can be replaced by the corresponding components in mice, leading to differences in the biological properties of the original tumor.

In view of this imperfection, we developed an optimized drug selection model based on the Alphacait screening system that combines artificial intelligence, synthetic lethal and combinational chemistry, which allows rapid selection of candidates from millions of drug combinations. We want to provide physicians with individualized drug therapy through a new in vitro and in vivo drug-sensitive screening technique, to achieve rapid and accurate selection of cancer clinical treatment.

In order to achieve the two key requirements of tumor tissue culture system in vitro, the establishment of tumor microenvironment we introduced the millimeter-sized microbeads, based on combinatorial chemistry in the culture medium. The surface of the microbeads is coated with small molecules that can specifically absorb high levels of metabolites secreted by the tumor cells into the matrix, thereby mimicking in vivo circumstances. In short, we innovatively applied microbeads technology to solve the inherent limitations of 3D organoid culture - no blood circulation in vitro.

Purpose and design Primary endpoint: progression-free survival (PFS) Secondary endpoints: overall survival (OS); disease control rate (DCR), objective response rate (ORR); safety; blood test and gene test in the aspect of biomarkers. Expectations of exploratory markers for this study include the status of exploratory biomarkers associated with immunohistochemistry (IHC) or quantitative reverse transcription polymerase chain reaction (qRT-PCR), a new generation sequencing method (NGS), Nanostring technique and / or other methods to evaluate archived and/or newly acquired tumor tissue, as well as its association with disease status and/or (Including but not limited to somatic mutations and other exploratory markers) according to qRT-PCR and NGS techniques, and to evaluate the relationship between the therapeutic response, the status of the biomarker during exploratory treatment and during treatment, and the evaluation of plasma, serum or whole blood samples (including but not limited to somatic mutations and other exploratory markers) The association of the above markers with disease status and / or therapeutic response.

Research design This is a single-center, open-label, single-arm, non-randomized study designed to evaluate PFS, safety, overall survival (OS), objective response rate (OPR), disease control rate (DCR) and biomarkers of cancer therapy based on the Alphacait screening system in subjects with advanced malignant tumor.

List of drugs used by the Alphacait screening system is as follow:

Non chemotherapy drug

Albendazole Tablets, Alfacalcidol Soft Capsules, Aripiprazole Tablets, Anastrozole Tablets, Azithromycin, Acyclovir Dispersible Tablets, Aztreonam, OLanzapine Tablets, Omeprazole Enteric-coated Capsules, Ornidazole and Sodium Chloride Injection, resveratrol, citicoline sodium injection, Bevacizumab，Avastin, Phenobarbital, Amlodipine Besylate Tablets, phenytoin sodium tablet, Piroxicam tablets, Allopurinol tablets, Propylthiouracil Tablets, Sodium Valproate for Injection, Nuprin Tablets, Goserelin Acetate Sustained-Release Depot, Zoladex, Megestrol Acetate Dispersible Tablets, Prednisone Acetate Tablets, Desmopressin Acetate Injection, Low-molecular-weight Heparin Sodium Injection, Digoxin Tablets, Dexamethasone Sodium phosphate Injection, Bacillus Licheniformis Capsule, tabellae paracetamol, Levodopa and Benserazide Hydrochloride Tablets, Domperidone Tablets, Metformin, Famotidine tablets, Fenbendazole, Nitrofurantoin Enteric-coated Tablets, Fluconazole and Sodium Chloride Injection, Haloperidol Injection, Flupentixol and Melitracen Tablets, Compound Zedoary Turmeric Oil Suppositories, Compound Sulfamethoxazole Injection, Compound Hypotensive Tablets, Bisoprolol Fumarate Tablets, Quetiapine Fumarate Tablets, Injection Mannitou, Heparin sodium, Bismuth Potassium Citrate Tablets, Banan tablet, Erythromycin enteric capsules, Metoprolol succinate sustained-release tablets, Warevan tablet, Huaier granule, Cyclosporine, Progesterone injection, Gabapentin capsules, Mebendazole Chewable Tablets, Apatinib Mesylate, Phentolamine Mesylate Injection, Imatinib Mesylate, Neostigmine Methylsulfate Injection, Imatinib Mesylate Tablets, Thiamazole Tablets, Metronidazole, Colloidal Bismuth Pectin Capsules, Metoprolol Tartrate Tablets, Carbamazepine Tablets, Captopril Tablets, Clarithromycin Sustained-release Tablets, Clindamycin Phosphate Injection, Lamictal, Letrozole Tablets, Lara chips, Tripterygium Glycosides, Atorvastatin, Ribavirin injection, Rifampicin Capsules, Risperidone Tablets, Primaquine Diphosphate, Chloroquine Phosphate Tablets, Amikacin Sulfate Injection, Atropine sulphate injection, Magnesium sulfate injection, Azathioprine Tablets, Sulfasalazine Enteric-coated Tablets, Roxithromycin Soft Capsules, Clozapine Tablets, Desloratadine Tablets, Flupirtine Maleate, Fluvoxamine Maleate Tablets, Chlorphenamine Maleate Tablets, Enalapril Maleate Tablets, Meloxicam, Mesalazine Enteric-coated Tablets, Mirtazapine, Naproxen Tablets, Nikethamide Injection, Nimodipine Injection, Nitrendipine Tablets, Norfloxacin Capsules, Hydroxycarbamide Tablets, Artemisinin, Benzylpenicillin sodium, Hydrocortisone Injection, Citalopram Hydrobromide Tablets, Gentamicin, Colchicine Tablets, Doxifluridine Capsules, Deslanoside Injection, Ciprofloxacin Lactate and Sodium Chloride Injection, Celecoxib Capsules, Trifluoperazine, Tetrastigma hemsleyanum Diels et Gilg, Thalidomide Tablets, Sulpiride Tablets, Diclofenac Potassium Capsules, Clostridium butyricum TO-A, Dihydroartemisinin and Piperaquine Phosphate Tablets, Tetracycline Tablets, Lithium Carbonate Sustained-release Tablets, Tegafur Injection, Teicoplanin, Tinidazole and Sodium Chloride Injection, Cefoxitin, Ceftizoxime Sodium, Topiramate Tablets, Vancomycin, Tretinoin Tablets, Vemurafenib, Vitamin A, Vitamin B2 Tablets, Vitamin D2 Injection, Cimetidine Tablets, Cimetidine Injection, Nifedipine Sustained Release Tablets, Nitroglycerin Injection, Isosorbide Dinitrate Injection, Valsartan Dispersible Tablets, Simvastatin Tablets, Thymalfasin, Ursodeoxycholic Acid, Folic acid calcium salt hydrate, Amitriptyline Hydrochloride Tablets, Bupropion Hydrochloride Sustained-Release Tablets, Amiodarone Hydrochloride Tablets, Ondansetron Hydrochloride Injection, Betahistine Hydrochloride Injection, Diphenhydramine Hydrochloride Injection, Bupropion Hydrochloride Injection Tablets, 3-Hydroxytyramine hydrochloride, Doxepin Hydrochloride, Flunayizine Hydrochloride Capsules, Prozac, Metoclopramide Dihydrochloride Injection, Arginine Hydrochloride Injection, Clindamycin Hydrochloride Injection, Raloxifene Hydrochloride Tablets, Ranitidine Hydrochloride Capsules, Lidocaine Hydrochloride Injection, Lobeline Hydrochloride Injection,, Chlorpromazine, Clomipramine Hydrochloride Tablets, Omeprazole Magnesium Enteric-coated Tablets, Mexiletine Hydrochloride Tablets, Paroxetine Hydrochloride Tablets, Procaine Hydrochloride for Injection, Trazodone Hydrochloride Tablets, Daunorubicin hydrochloride, Cyproheptadine Hydrochloride Tablets, Sertraline Hydrochloride Tablets, Tamsulosin Hydrochloride Sustained Release Capsules, Terazosin Hydrochloride Tablets, Verapamil Hydrochloride Tablets, Venlafaxine Hydrochloride Capsules, Raceanisodamine Hydrochloride Injection, Berberine Hydrochloride Tablets, Ethambutol Hydrochloride Tablets, Levofloxacin Hydrochloride for Injection, Itraconazole, Ivermectin, IPTG；Isopropyl-β-D-thiogalactoside, Isopropyl-beta-D-thiogalactopyranoside, Isoniazid Tablets, Indapamide Tablets, Indomethacin Enteric-coated Tablets, Amoxicillin Sodium and Clavulanate Potassium for injection, Azithromycin for Injection, Acyclovir for Injection, Ampicillin Sodium Injection, Omeprazole Sodium for Injection, Oxacillin Sodium for Injection, Biapenem for Injection, Benzathine Penicillin For Injection, Sodium Valproate for Injection, Ganciclovir, Fosfomycin Sodium for Injection, Asparaginase, Urokinase for Injection, Piperacillin Sodium for Injection, Artesunate for Injection, Sodium Nitroprusside, Diltiazem Hydrochloride for Injection, Recombinant Human Interferon gamma for Injection, Levobupivacaine, Levothyroxine Sodium Tablets, Levofloxacin Tablets

Chemotherapy and target therapy drugs

Aidi injection, Oxaliplatin for Injection, Epirubicin, Dacarbazine, Dabrafenib, mesylate, Dabratinib, Dasatinib Tablets, Sorafenib Tosylate Tablets, Doxorubicin, Docetaxel, 5-Fluorouracil, Juyuansuan Tamoxifen, Cino bufotalin, Cyclophosphamide, Gefitinib (pure) powder, Gemcitabine hydrochloride, Methotrexate, Carboplatin, Capecitabine, Kanglaite Injection, Raltitrexed, Mabthera, Lobaplatin for Injection, Mitoxantrone, Nedaplatin, Mercaptopurine, Cisplatin, Mitomycin for Injection, Tacrolimus, Tegafur, Gimeracil and Oteracil Potassium, Temozolomide, Cetuximab Solution for Infusion, Lobaplatin for Injection, Mitoxantrone, Nedaplatin, Mercaptopurine, Cisplatin, Mitomycin for Injection, Tacrolimus, Tegafur, Gimeracil and Oteracil Potassium, Temozolomide, Cetuximab Solution for Infusion

Chinese Herb Medicine

English Name Latin Name Job's tears seed Coicis Semen, Japanese Ardisia Herb Japanese Ardisia Herb, White Hyacinth Bean Semen Dolichoris Album, Spreading Hedyotis Herb Hedyotis diffusa, Willowleaf Swallowwort Rhizome Rhizoma Cynanchi Stauntonii, Large head Atractylodes Rh Rhizoma Atractylodis Macrocephalae, Sessile Stemona Root Japanese Stemona Root, Lily Lilium brownii var. viridulum, Seman Platycladi Seman, Isatis root Isatis tinctoria, Herba Lobeliae Chinensis Lobelia chinensis Lour, Pinellia ternata Pinellia ternata (Thunb.) Breit, Scutellaria barbata Scutellaria barbata, CoasiaI GIehnia Root Glehnia littoralis, Fritillary fritillary, Ficus pumila Linn Ficus pumila, Seed-coat of Hyacinth Dolichos, Areca Seed, Betel Nut Semen Arecae, Malaytea Scurfpea Fruit Fructus Psoraleae, Semen raphani , Silkworm shit Faeces Bombycis, Siberian Cocklour Fruit Fructus Xanthii, Rhizome of Swordlike Atractylodes Rhizoma Atractylodis, Root of Chinese Thorowax Radix Bupleuri, Radices paeoniae rubra Paeoniae Rubra Radix, Dan - shen Root Salviae Miltiorrhizae Radix, Tree Peony Root - bark Moutan Radicis Cortex, Chinese Goldthread Rhizome Coptidis Rhizoma, Skunk Bugbane Rhizome Cimicifugae Foetidae Rhizoma, Coix seed Semen Coicis Szechwan Chinaberry Fruit Fructus Meliae Toosendan, Radix Cyathulate Radix Cyathulae, Common Andrographis Herb Herba Andrographis, Radix et Caulis Acanthopanacis Senticosi Radix et Caulis Acanthopanacis Senticosi, Japanese Thistle Herbor Root Herba seu Radix Cirsii Japonici, Indigowoad Leaf, Leaf of Indigowoad Folium Isatidis, Danshen Root, Root of Dan-shen Salviae Miltiorrhizae Radix et Rhizoma, Root of Pilose Asiabell Radix Codonopsis, Fructus Oryzae Germinatus Fructus Oryzae Germinatus, Humifuse Euphorbia Herb Herba Euphorbiae Humifusae, Chinese Waxgourd Peel Exocarpium Benincasae, Waxgourd seed Semen Benincasae, Rabdosia rubesens,hamst Rabdosia rubescens, Rhioxma Curcumae Aeruginosae Rhizoma Curcumae, Divaricate Saposhnikovia RootRadix Saposhnikoviae, Indian Buead Poria, Pine among the Indian Bread, Blighted Wheat Fructus Tritici Levis, Radix Glycyrrhizae Radix Glycyrrhizae, Toad skin, Perfoliate Knotweed Herb Polygonum perfoliatum, Ligusticum sinense Oliv Rhizoma Ligustici, Barbary Wolfberry Fruit Fructus Lycii, Herba Pogostemonis Herba Pogostemonis, Sargassum Sargassum, Yerbadetajo Herb Herba Ecliptae Eclipta prostrala, Terminalia chebula Retz, Taxus chinensis Taxus chinensis (Pilger) Rehd, Flos Carthami Flos Carthami, Root of Kirilow Rhodiola Herba Rhodiolae, Figwortflower Picrorhiza Rhizome Rhizoma Picrorhizae, Polygonum cuspidatum Rhizoma Polygoni Cuspidati, Pricklyash Peel Pericarpium Zanthoxyli, Talcum Talcum, Exocarpium Citri Grandis Exocarpium Citri Grandis, Phellodendron Chinese Schneid Cortex Phellodendri, Manyflower Solomonseal Rhizome Rhizoma Polygonati, Radix Astragali Radix Astragali seu Hedysari, Radix Scutellariae, Flos Celosiae Cristae Flos Celosiae Cristatae, Suberect Spatholobus Stem Caulis Spatholobi, Rhizoma Curcumae Longae Rhizoma Curcumae Longae, Christina Loosestrife HerbHerba Lysimachiae, Japanese Honysuckle Flower Bud Flos Lonicerae, Cherokee Rose Fruit Fructus Rosae Laevigatae, Chrysanthemum flower Flos Chrysanthemi, Spikemoss Herba Selaginellae, Cassia seed Semen Cassiae, Lightyellow sophora root Radix Sophorae Flavescentis, Kelp Laminariae Thallus, Semen Litchi Semen Litchi, Chinese trumpet creeper Campsis grandiflora, Diverse Wormwood Herb Herba Artemisiae Anomalae, Radix Gentianae Gentiana Scabra Bunge, Reed Rhizome Stemmacanthae Unifori Radix, Caulis Trachelospermi Trachelospermi Jasminoidis Caulis, Lv Bean Spermodermis Phaseoli Radiati, European Verbena Herb Herba Verbenae Officinalis, Herba Portulacae Portulaca oleracea L, Radix Ophiopogonis Ophiopogonis Radix, Fructus Hordei Germinatus Hordei Germinatus Fructus, Concha Ostreae Concha Ostreae, Costustoot, Common Vladimiria Root Aucklandiae Radix, Fructus Ligustri Lucidi Ligustri Lucidi Fructus, Fortune Eupatorium Herb Eupatorii Fortunei Herba, Folium Eriobotryae Eriobotryae Japonicae Folium, Dandelion Herba Taraxaci, Flower of Shepherdspurse Capsella bursa-pastoris (L.)Medic), Rhizoma Homalomenae Rhizoma Homalomenae, Gordon Enryale Seed Euryales Semen, Radix Gentinae Gentianae Macrophyllae Radix, Cortex Fraxini Fraxini Cortex, Caulis SinomeniiI Caulis Sinomenii, Semen Celosiae Celosiae Argenteae Semen, Herba Dianthi Dianthi Superbi Herba, Caulis Lonicerae Lonicerae Caulis, Cortex CinnamoniCinnamomi Cassiae Cortex, Rhizoma Srarganii Rhizoma Sparganii, Sanchi Panax pseudo-ginseng var, Radix tetrastigme Tetrastigma hemsleyanum Diels et Gilg, Folium Mori Mori Folium, Chinese yam Dioscorea opposite, Amorphophallus rivieri Durieu Amorphophallus rivieri Durieu, Snake venom, Snake Slough Serpentis Periostracum, Rhizoma Belamcandae rhizoma belamcandae, Largetrifoliolious Bugbane RhizmomeRhizoma Cimicifugae, Radix Sanguisorbae SanguisorbaofficinalisL, Eucommia ulmoides Oliver Eucommia ulmoides, Rhizoma Zingiberis RecensZingiber officinale Roscoe, Salvia chinensis Benth Salvia chinensis Benth, Folium Photiniae Photinia serrulata Lindl, Lignum Sappan Lignum Sappan, Semen Persicae Semen Persicae, Radix Asparagi Radix Asparagi, Root of Nakedcaule Groundsel Radix Semiaquilegiae, Root of Common carpesium Herba Carpesii Abrotanoidis, Semen lepidii Semen Lepidii, Herb of Tuberculate Speranskia Phryma leptostachya L. subsp. asiatica (Hara), China Dodder Semen Cuscutae, Semen Vaccariae Semen Vaccariae, Herb of Coffee Senna Cassia occidentalis Linn, Fructus Mume Fructus Mume, Root of Combined Spicebush Radix Linderae, Fig Ficus carica Linn, Medicinal Evodia Fruit Evodia rutaecarpa (Juss.) Benth, Chinese Gall, Chinese Nut-gall Rhus chinensis Mill, Sessileflower Acanthopanax Bark Cortex Acanthopanax Radicis, All-grass of Bluecalyx Japanese Rabdosia, Fructus Foeniculi Fructus Foeniculi, Common Cephalanoplos Herb Cirsium setosum (Willd.) MB, Flos Magnoliae Flos Magnoliae, Paniculate Swallowwort Root Cynanchum paniculatum (Bunge) Kitagawa, Linseed,seed of Flax Linseed seed of Flax, Fructus Alpiniae Oxyphyllae Alpinia oxyphylla Miq, Job's tears seed Semen Coicis, Herba Artemisiae Scopariae ArtemisiacapillarisThunb, Folium Ginkgo Ginkgobiloba, Heartleaf Houttuymia Herb Houttuynia cordata Thunb, Turmeric Root-tuber Radix Curcumae, Akebia Fruit Foreknowledge, Hiraute Shiny Bugleweek Herb Aconitum gymnandrum Maxim, Rhizoma Paridis RhizomaParidis, Polyporus Polyporus, Root of Sinkiang Arnebia Lithospermum erythrorhizon Sieb. et Zucc, Herba Violae Viola yedoensis Makino, Fluoritum Fluoritum Caulis Perillae Perilla frutescens （L.）Britton

ELIGIBILITY:
Inclusion Criteria:

1. Advanced recurrent or metastatic malignant tumor confirmed by pathological diagnosis;
2. At least one measurable malignant lesion;
3. Failed previous standard treatment or with tumor recurrence, and no standard therapeutic regimen available;
4. No radiation therapy within last four weeks or recovered from last radiation related acute complication, if applicable; prophylactic brain radiation therapy or palliative radiation treatment for bone metastasis is acceptable;
5. No gender requirement and must be no younger than18 years old;
6. ECOG PS: score 0-2;
7. Life expectancy more than three months;
8. Patient's organ function level should meet these criteria:

(1) CBC should meet these criteria: ANC≥1.5×109 /L，PLT≥100×109/L，Hb≥ 100 g/L; (2) Chemistry should meet these criteria: TBIL<1.5×ULN，ALT、AST< 2.5×ULN（if with liver metastasis ALT、AST<5×ULN） BUN and Cr ≤1×ULN or Cr clearance ≥50ml/min（Cockcroft-Gault formula） 9. Agree to use appropriate contraceptive measure during the study period and until 8 weeks after the last study drug is given. Or patient has been surgically sterilized.

10. Qualified candidate should voluntarily participate this study, sign informed consent forms and be compliant with the study protocols and follow-up visit(s).

Exclusion Criteria:

1. Symptomatic brain metastasis (could still enroll into the study if treatment finished 21 days prior to the enrollment and the patient is stable, but brain MRI, CT or angiogram is needed to rule out no intracranial hemorrhage)
2. Following cardiac disease: second-degree or above cardiac ischemia or myocardial infarction, uncontrolled arrhythmias (including QTc interval male>450 ms, female>470ms), according to NYHA criteria, III to IV cardiac insufficiency, or echocardiogram reveals left ventricular ejection fraction (LVEF) <50%;
3. History of pulmonary interstitial lung disease or active interstitial lung disease;
4. Coagulation dysfunction (INR >1.5 or PT>ULN+ 4sec, or PTT>1.5 ULN), with bleeding tendency or currently receiving thrombolysis therapy or anticoagulation treatment;
5. Clinical bleeding episode or bleeding tendency within past three months, such as GI bleeding, hemorrhagic gastric ulcer, stool guaiac++ positive, or with vasculitis；
6. Arterial or venous thrombosis within last 12 months, such as various types of CVA, DVT or PE patients;
7. Known hereditary or acquired bleeding or hypercoagulable state (such as hemophilia, coagulating dysfunction, thrombocytopenia, hypersplenism);
8. Major surgery, trauma, fracture or ulcer within past 4 weeks;
9. Active infection requiring antibiotics, antifungal or antiviral treatment;
10. Patient has a history of psychiatric medication abuse and cannot be abstinent from the psychiatric medication, or with mental disorder;
11. Participation of other cancer chemotherapy clinical study within past 4 weeks;
12. History of uncured coexisting cancer, no including cured basal cell carcinoma, cervical cancer in situ, or superficial bladder cancer;
13. Pregnant or breast feeding women; fertile patients no willing or able to take effective contraceptive measures;
14. Any circumstances that might affect the proceeding of the clinical trial and/or research result analysis, as determined by the clinical investigator(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 36 months
  Progression-free survival (PFS) is defined as the time from assignment in the trial to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival(OS) | 36 months
  Defined as the time from assignment to death from any cause.
Overall response rate (ORR) | 36 months
  Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy
Disease control rate(DCR) | 36 months
  Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response or stable disease to therapy
Incidence of Treatment-Emergent Adverse Events | 36 months
  Drug-related adverse reactions must be recorded, mainly in the following：myelosuppression including neutropenia, anemia and thrombocytopenia;Cardiac toxicity; muscle fatigue, pain, imbalance; Oral ulcers: the patient's gums, cheeks, throat and tongue are prone to ulcers;nausea, vomiting, constipation or diarrhea;hair loss;skin discomfort;hormonal fluctuations, sexual dysfunction, infertility; damage of the kidney;anxiety and depression.
Biomarkers | 36months
  Expectations of exploratory markers for this study include the status of exploratory biomarkers associated with immunohistochemistry (IHC) or quantitative reverse transcription polymerase chain reaction (qRT-PCR), a new generation sequencing method (NGS), Nanostring technique and / or other methods to evaluate archived and/or newly acquired tumor tissue, as well as its association with disease status and/or (Including but not limited to somatic mutations and other exploratory markers) according to qRT-PCR and NGS techniques, and to evaluate the relationship between the therapeutic response, the status of the biomarker during exploratory treatment and during treatment, and the evaluation of plasma, serum or whole blood samples (including but not limited to somatic mutations and other exploratory markers) The association of the above markers with disease status and / or therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Haizhou Lou, MD, Principal Investigator — Sir Run Run Shaw Hospital; Linghua Zhu, MD, Principal Investigator — Sir Run Run Shaw Hospital; Enguo Chen, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, affiliated with Zhejiang University School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Through publication after study completion
Supporting Information: Study Protocol
Time Frame: 12/31/2018